CLINICAL TRIAL: NCT07036952
Title: Effect of Omega-3 Supplementation as Add on Therapy on Metabolic Syndrome in Women With Polycystic Ovary Syndrome: A Randomized Double-Blind, Placebo-Controlled Trial
Brief Title: Effect of Omega-3 Supplementation as Add on Therapy on Metabolic Syndrome in Women With Polycystic Ovary Syndrome.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Principal Investigator, Dr. Fariba kabir, Principal investigator: Dr. Fariba Kabir, MD, Bangabandhu Sheikh Mujib Medical University, Dhaka Bangladesh., Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BSMMU/2025/3950
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: PCOS (Polycystic Ovary Syndrome)
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Fatty Acids, Omega-3; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 (Experimental): Participants received Omega-3 1gm tablet orally twice daily for 12 weeks.
  Interventions: Drug: Omega 3 fatty acids; Drug: Omega -3 fatty acids
- placebo (Placebo Comparator): Participants received Omega-3 1gm placebo matching Omega-3 tablet orally twice daily for 12 weeks
  Interventions: Drug: Omega 3 fatty acids; Drug: Omega -3 fatty acids

INTERVENTIONS:
Drug: Omega 3 fatty acids — 1gm tab twice daily.
Drug: Omega -3 fatty acids — 1gm tablet twice daily.

SUMMARY:
The goal of this clinical trial is to learn if Omega-3 works to treat Polycystic ovary syndrome in women. It will also learn about the safety of drug Omega-3. The main questions it aims to answer are:

Does Omega-3 lower the number of times participant to treat metabolic syndrome What medical problems do participants have when taking drug Omega-3.Researchers will compare drug Omega-3 to a placebo (a look-alike substance that contains no drug) to see if drug Omega-3 used to treat PCOS.

Participants will:

Take Omega-3 or a placebo every day for 3 months Visit the clinic once every 6 weeks for checkups and tests Keep a diary of their symptoms and menstrual history.

DETAILED DESCRIPTION:
This research will be a single center study, utilizing a double-blind, randomized placebo-controlled trial design. A total of 62 women, with newly diagnosed PCOS, age range from 18-36 years will randomly be assigned to receive either Omega-3 supplementation (1gm twice daily) or a placebo for 12 weeks. Biochemical and anthropometric measurements, including lipid profile, fasting blood sugar, blood pressure, inflammatory markers (CRP) and body composition such as BMI, waist circumference will be assessed at baseline and post-intervention. Follow-up assessments will be conducted three months after supplementation to evaluate the sustainability of metabolic changes. For independent samples; t-test will be utilized to analyze the average differences in metabolic biomarker levels between the group receiving Omega-3 supplements and the group receiving a placebo. The Chi-square test or Fisher's exact test will be employed to compare the percentage of participants may show a significant change in metabolic biomarker in the group that received Omega-3 versus the group that received a placebo. Pearson or Spearman correlation tests will be used to explore any relationships between baseline Omega-3 levels and baseline inflammatory marker (CRP) and lipid profile levels, as well as between the change in Omega-3 levels and the change in inflammatory marker (CRP) and lipid profile levels

ELIGIBILITY:
Inclusion Criteria:• Rotterdam criteria for PCOS (Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS) 2004).

* Age above 18 years up to 35 years
* Newly diagnosed case of PCOS.

Exclusion Criteria:• Pregnancy and lactating mother.

* History of diabetes mellitus (except those meeting metabolic syndrome criteria)
* Any chronic illness (e.g. liver disease, kidney disease, cardiovascular disease)
* Any acute or chronic infective or inflammatory disease.
* Patients receiving Omega-3 supplementation within the last three months.
* Exclusion of PCOS mimicking disease include hyperprolactinemia, adrenal hyperandrogenism, ovarian hyperandrogenism, cushing's syndrome, acromegaly etc.
* Known allergy to fish oil or Omega-3 supplements.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female age range:18-36 years
Enrollment: 68 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Effect of Omega-3 Supplementation as Add on Therapy on Metabolic Syndrome in Women with Polycystic Ovary Syndrome: A Randomized, Double-Blind, Placebo-Controlled Trial | 12 weeks.
  Changes in Lipid profile (Triglycerides, HDL-Cholesterol) Omega3 reduce Triglyceride and increase HDL Cholesterol Changes in CRP Plasma Omega-3 level (changes in plasma DHA and EPA conc. from baseline to 12 weeks) Changes in BMI,Omega3 reduce weight as well as BMI. Improvement of menstrual cycle regularity. Improvement of hirsutism.

CONTACTS AND LOCATIONS:
Locations (1):
- Fariba kabir, Dhaka, Bsmmu, Bangladesh

IPD SHARING:
Plan to Share IPD: No